CLINICAL TRIAL: NCT07209085
Title: SPARC: A Prospective, Multicenter Evaluation of the Safety and Performance of the Artero Intravascular Lithotripsy System for the Treatment of Peripheral Artery Disease and Remodeling Arterial Calcium
Brief Title: A Study to Evaluate the Safety and Effectiveness of the FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System in Adults With Peripheral Artery Disease (PAD)
Acronym: SPARC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FastWave Medical (Industry)
Collaborators: Rede Optimus Hospitalar SA (Network); Medical Metrics Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FW100206/ Rev A
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Artery Disease (PAD)
Keywords: Peripheral Artery Disease (PAD); Lower Extremity Arterial Disease; Femoropopliteal Artery; Arterial Calcification; Vascular Calcification; Endovascular Therapy; Intravascular Lithotripsy (IVL); FastWave Artero IVL System; Angioplasty
MeSH Terms: conditions — Peripheral Arterial Disease; Vascular Calcification

STUDY DESIGN:
Intervention Model Description: Single-arm pivotal study evaluating the FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System in subjects with femoropopliteal arterial disease and moderate to severe calcification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Experimental: FastWave Artero™ IVL System (Experimental): All participants in this single-arm study will receive treatment with the FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System during a single endovascular index procedure performed to open blocked femoropopliteal arteries that contain moderate to severe calcium buildup.
  The IVL System includes a generator and a balloon-based catheter that delivers short bursts of pulsatile sonic pressure waves inside the artery to fracture calcium within the vessel wall. This improves vessel flexibility and allows dilation at low balloon pressures to restore blood flow.
  During the index procedure, investigators may perform multiple balloon inflations or treatment cycles as needed to treat the full length of the target lesion. Adjunctive therapies, such as balloon angioplasty or stent placement, may be used at the investigator's discretion to achieve optimal vessel opening.
  Interventions: Device: FastWave Artero™ Peripheral IVL System

INTERVENTIONS:
Device: FastWave Artero™ Peripheral IVL System — The FastWave Artero™ Peripheral IVL System includes a generator and a balloon-based catheter designed to treat calcified blockages in peripheral arteries. During a single endovascular index procedure, the catheter is positioned within the target femoropopliteal artery and inflated at low pressure. The device emits short bursts of pulsatile sonic pressure waves that fracture calcium deposits, improving vessel flexibility and allowing dilation at low balloon pressures to restore blood flow. Multiple inflations may be performed as needed. Adjunctive angioplasty or stenting may be used at the investigator's discretion.
  Other Names: FastWave Artero IVL Catheter; Intravascular Lithotripsy System

SUMMARY:
The purpose of this clinical study is to learn if the FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System is safe and works well to help people with peripheral artery disease (PAD) who have hard, calcium-filled blockages in their leg arteries.

The study will test the idea that using sound waves inside the artery can safely break up calcium and make it easier to open the artery so blood can flow better.

The main question this study is trying to answer is:

Can treatment with the FastWave Artero™ IVL System safely widen blocked leg arteries and lower the chance of serious problems during or after the procedure?

About 110 adults at up to 30 medical centers in the United States will take part. Everyone in the study will receive the IVL treatment.

During the study, participants will:

Have a minimally invasive procedure using the FastWave IVL System

Stay for a short observation period after the procedure

Return for follow-up visits about 30 days and 6 months later

Researchers will look at how well the arteries open, how long they stay open, and whether any major complications occur. The results will help determine if the FastWave Artero™ IVL System can be used as a safe and effective treatment for people with PAD and severe calcium buildup in the leg arteries.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) happens when plaque and calcium build up inside the arteries of the legs. This buildup narrows the arteries and limits blood flow, which can cause pain, limited mobility, and slow healing of wounds. Treating arteries that contain a large amount of calcium can be difficult because the calcium makes the artery wall stiff and hard to open with standard balloons or stents.

The FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System is designed to improve treatment for people with moderate to severe calcium in their leg arteries. The system includes a generator and a small balloon catheter that emits short bursts of sound energy (lithotripsy). These sound waves gently fracture calcium deposits while protecting the softer tissue of the artery. After the calcium is cracked, the artery can be widened using low balloon pressure, which may help blood flow more easily and lower the risk of tearing or other damage.

This prospective, multi-center, single-arm clinical study will evaluate the safety and effectiveness of the FastWave Artero™ IVL System in adults with PAD who have calcified blockages in the femoral or popliteal arteries. The study will enroll up to 110 participants at as many as 30 U.S. investigational sites. All participants will receive the FastWave IVL treatment during a standard minimally invasive endovascular procedure.

The primary safety endpoint is the proportion of participants free from major adverse events (such as serious vessel injury, emergency surgery, or unplanned major amputation) through 30 days after the procedure.

The primary effectiveness endpoint is successful treatment of the blocked artery, defined as less than 50 percent narrowing remaining after IVL, with or without the use of additional devices.

Secondary assessments will include degree of residual narrowing (≤30%), use of adjunctive therapies, and improvements in vessel patency and clinical symptoms through 6 months. These data will also be used to compare outcomes to a historical performance goal based on prior intravascular lithotripsy studies in peripheral arteries.

Participants will be followed at discharge, 30 days, and 6 months to assess safety, vessel imaging, and symptom changes. A small number of sites will also participate in an optional intravascular ultrasound (IVUS) sub-study to collect detailed imaging data on how the FastWave device interacts with the artery wall.

Findings from this pivotal study are intended to support a future U.S. Food and Drug Administration (FDA) 510(k) submission for the FastWave Artero™ Peripheral IVL System as a treatment for calcified peripheral arterial disease.

ELIGIBILITY:
Inclusion Criteria

1. Subject is able and willing to comply with all assessments in the study.
2. Subject or subject's legal representative has been informed of the nature of the study, agrees to participate, and has signed the approved consent form.
3. Subject is ≥ 18 years of age.
4. Rutherford Clinical Category 2, 3 or 4
5. Resting ABI of ≤0.90, or ≤0.75 after exercise, of the target leg.
6. Lesion calcification is moderate or severe using the PARC3calcium classification definition, or by intravascular ultrasound (IVUS) determined by the investigator.

   1. Moderate is defined as ≥ 180º to 270º and < 50% of the total lesion length.
   2. Severe is defined as >270º and > than 50% of the total lesion length.
7. Estimated life expectancy >1 year, in the opinion of the investigator at the time of enrollment.
8. Target lesion that is in a native de novo femoral-popliteal arteries. Non-target lesions can be in the iliac arteries (inflow).
9. The subject is a suitable candidate for angiography and endovascular intervention, in the investigator's opinion or per the hospital guidelines.
10. In the opinion of the investigator by visual estimate, the target lesion is ≥70% stenosis or is occluded.
11. According to the visual estimate, the target lesion reference vessel diameter is between 3.5mm and 8.0mm.
12. The total planned target lesion length must be ≤220 mm.

    1. Tandem lesions (i.e., two or more lesions in close proximity) may be considered a single lesion if the distance between them is ≤ 30 mm.
    2. Multiple target vessel beds and discrete (non-contiguous) lesions may be treated, provided the combined total length of all treated lesions does not exceed 220 mm.
13. Subject has at least one patent tibial vessel on the target leg with runoff to the foot, defined as no stenosis >50% distal to the target lesion.

    a. If the peroneal artery, at least one collateral must supply the foot.
14. Retrograde access is permitted for lesion crossing; however, the FastWave Artero™ Peripheral Intravascular Lithotripsy (IVL) System must be deployed from antegrade (either ipsilateral or contralateral) access.

Exclusion Criteria

1. Planned use of atherectomy, scoring or cutting balloons, or any investigational device other than lithotripsy.
2. Rutherford Clinical Categories 0, 1, 5, and 6.
3. The investigator determined no or mild calcium in the target lesion.
4. Subject has outflow disease in which no tibial vessel has <50% stenosis. Staged or concomitant intervention to the tibial vessels is not allowed.
5. The subject has significant inflow disease, defined as >50% stenosis or occlusion in the inflow tract proximal to the target lesion, that has not been successfully treated prior to treatment of the superficial femoral artery (SFA) or popliteal lesion.

   a. Successful treatment is defined as residual stenosis ≤30% without a flow-limiting dissection or vessel perforation.
6. The subject has significant outflow disease in which no tibial vessel has <50% stenosis. Staged or concomitant intervention to the tibial vessel is not allowed.
7. Inability to pass the guidewire across the target lesion.
8. In-stent restenosis within the lesion(s) to be treated.
9. Lesions within autologous or synthetic vessel grafts.
10. Evidence of aneurysm or thrombus in the vessels to be treated.
11. History of prior endovascular or surgical intervention on the index limb within 14 days prior to the index procedure, unless part of a pre-specified, staged treatment plan.
12. Intervention on the contralateral limb is required within the next 14 days.
13. History of thrombolytic therapy within two weeks of enrollment.
14. Subject has a known hypercoagulable state, coagulopathy, or has a bleeding diathesis, thrombocytopenia with platelet counts less than 100,000/microliter, or International Normalized Ratio (INR) >1.5.
15. Subject in whom antiplatelet or anticoagulant therapy is contraindicated.
16. Myocardial infarction within 60 days prior to enrollment.
17. History of stroke within 60 days prior to enrollment.
18. History of unstable coronary artery disease or other uncontrollable comorbidity resulting in hospitalization within the last 60 days prior to enrollment.
19. Subject has acute or chronic renal disease defined as serum creatinine of >2.5 mg/dL or >220 µmol/L, or on dialysis.
20. Subject has an active infection requiring antibiotic therapy.
21. Subject has known allergy to contrast agents, medications, or catheter materials used to perform endovascular intervention that cannot be adequately pre-treated.
22. Subject is pregnant or nursing.
23. Subject is participating in another research study involving an investigational agent (pharmaceutical, biologic, or medical device) that has not reached the primary endpoint.
24. Subject has other medical, social, or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Procedural Success | Immediately Following the Index Procedure
  Procedural success is defined as ≤50% residual stenosis in the target lesion after treatment with the FastWave Artero™ IVL System, with or without adjunctive therapy (e.g., angioplasty or stenting).
Freedom from Major Adverse Events (MAE) at 30 Days | 30 Days Post-Procedure
  The percentage of subjects free from major adverse events (MAE) through 30 days following the index procedure. MAE is defined as unplanned surgical revascularization of the target limb, major amputation of the target limb, symptomatic thrombosis or embolism requiring intervention, vessel perforation requiring covered stent, or unresolved flow-limiting dissection.

SECONDARY OUTCOMES:
Residual Stenosis ≤30% | Immediately post-procedure
  The percentage of subjects achieving ≤30% residual stenosis in the target lesion as measured by angiography following treatment.
Incidence of Adjunctive Therapy | Immediately post-procedure
  The percentage of subjects requiring adjunctive therapy (angioplasty, stent placement, or other devices) to achieve procedural success.
Primary Patency | 30 days and 6 months post-procedure
  The percentage of target lesions maintaining primary patency, defined as freedom from clinically driven target lesion revascularization and duplex ultrasound evidence of ≤50% restenosis.
Freedom from Major Adverse Events (MAE) at 6 Months | 6 months post-procedure
  The percentage of subjects free from MAE through 6 months following the index procedure, using the same MAE definition as the primary safety endpoint.
Change in Ankle-Brachial Index (ABI) from Baseline | Baseline to 30 days and 6 months
  The Ankle-Brachial Index (ABI) is the ratio of ankle to arm systolic blood pressure. Scale range: 0.00-1.30 (values >1.30 indicate non-compressible arteries). Directionality: Higher ABI within the normal range indicates a better outcome (better limb perfusion); lower ABI indicates worse perfusion. If ABI is non-compressible (>1.30), Toe-Brachial Index (TBI) will be used per protocol.
Change in Rutherford Clinical Category (RCC) | Baseline to 30 days and 6 months
  Change in symptom severity using Rutherford Clinical Categories compared with baseline.
Change in Quality of Life (EQ-5D-5L) from Baseline | Baseline to 30 days and 6 months
  The EQ-5D-5L Index summarizes health across 5 domains with country-specific weights. Scale range (U.S. value set): -0.573 to 1.000. Directionality: Higher scores indicate a better outcome (better health status).
Change in Walking Impairment Questionnaire (WIQ) Scores from Baseline | Baseline to 30 days and 6 months
  The Walking Impairment Questionnaire (WIQ) assesses walking function across subscales (Distance, Speed, Stair-Climbing). Scale range (each subscale): 0 to 100. Directionality: Higher scores indicate a better outcome (less walking limitation/better function). Report each subscale separately.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared. Study results will be posted on ClinicalTrials.gov as required.